CLINICAL TRIAL: NCT04120272
Title: Discovery for Biomarkers and Risk Factors for Postoperative Delirium in Elderly Patients With Spine Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2019-0654
Record Dates: First submitted 2019-09-29; First posted 2019-10-09 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Spinal Disease
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gene expression and expression comparison in exosomes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delirium group: Group of patients with postoperative delirium
  Interventions: Procedure: Spine surgery
- Non delirium group: Group of patients without postoperative delirium
  Interventions: Procedure: Spine surgery

INTERVENTIONS:
Procedure: Spine surgery — Eligible Surgeries: lumbar spine fusion surgery, posterior cervical spine fusion surgery, or anterior cervical spine fusion surgery

SUMMARY:
Introduction: With the increase of the elderly population, the number of elderly patients undergoing surgery is increasing, and postoperative delirium is 11-51% depending on the type of surgery. In recent cohort studies have shown that delirium might reduce cognitive function and develop dementia.

Since delirium is difficult to treat, the key to treatment is prevention, and about 40% is prevented when prophylactic intervention is applied. However, delirium is difficult to diagnose and difficult to predict, therefore, biomarkers are needed to diagnose and prevention.

Exosome and brain efficiency test(electroencephalogram, and pulse wave test) have the potential of simple biomarkers that can diagnose postoperative delirium and predict cognitive decline.

Purpose: The purpose of this study is to investigate the risk factors affecting delirium in the elderly who have spinal surgery and to search for biomarkers of delirium for early detection and prevention of delirium.

DETAILED DESCRIPTION:
Method:

1. Study design: This study is a prospective investigation that identifies risk factors for postoperative delirium and searches for predictive biomarkers of delirium.
2. Inclusion criteria / Exclusion Criteria

   1. Inclusion criteria

      * Elderly patients over 70
      * Eligible Surgeries: lumbar spine fusion surgery, posterior cervical spine fusion surgery, or anterior cervical spine fusion surgery
   2. Exclusion Criteria

      * Patients with cognitive decline according to MMSE-DS outcome criterion
      * Patients diagnosed with malignant or benign tumors
      * If surgery is scheduled within 2 hours(micro surgery)
      * In case of difficulty in communication
      * History of brain neurological diseases (brain hemorrhage, stroke, dementia, Parkinson's, cognitive impairment diagnosis, etc.)
      * Patients diagnosed with alcoholism or drug addiction
      * Patients with surgical complications (post-operative bleeding, high fever over 39 degrees, etc.)
      * Patients undergoing re-operation due to surgery-related complications
3. Outcome

   1. Primary outcome: Urinary and Blood exosome, stool
   2. Secondary outcome: brain function test(electroencephalogram, pulse wave test, and cognitive test)
4. Measurement

   1. Delirium: Confusion Assessment Method(CAM), Korean-Delirium Rating Scale-R-98(K-DRS-R-98), Korean Nusing Delirium Scale(Nu-DESC)
   2. Cognitive function test: Mini-Mental State Examination-Dementia Screening(MMSE-DS), Montreal Cognitive Assessment(MoCA), Telephone interview for Cognitive Status(TICS)
   3. Depression: Geriatric Depression Scale Short Form Version (GDSSF-K)
   4. Activity Daily of Living: K-ADL, K-IADL
   5. Frail: Korean version of the FRAIL scale
   6. Nutrition: Mini Nutritional Assessment-Short Form
   7. patient-reported outcomes ; PROMIS-29

ELIGIBILITY:
Inclusion Criteria:

1. Elderly patients over 70
2. Eligible Surgeries: lumbar spine fusion surgery, posterior cervical spine fusion surgery, or anterior cervical spine fusion surgery

Exclusion Criteria:

1. Patients with cognitive decline according to MMSE-DS outcome criterion
2. Patients diagnosed with malignant or benign tumors
3. If surgery is scheduled within 2 hours(micro surgery)
4. In case of difficulty in communication
5. History of brain neurological diseases (brain hemorrhage, stroke, dementia, Parkinson's, cognitive impairment diagnosis, etc.)
6. Patients diagnosed with alcoholism or drug addiction
7. Patients with surgical complications (post-operative bleeding, high fever over 39 degrees, etc.)
8. Patients undergoing re-operation due to surgery-related complications

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Tertiary hospital, single institution
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-10-21 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Exosomes in Urine: Differences in Gene Expression | Just before surgery
  - Gene expression and expression comparison in exosomes The gene expression difference is determined using the SAM tool and DEseq2, and the Gene Ontology (GO) Database (www.geneontology.org) and the KEGG database (www.genome.jp/kegg) are used to find the correlation between gene functions.
  In the case of miRNA, there will be a regulatory function of the coding gene, so for this purpose, an integrative analysis is performed to identify the mRNA-miRNA interaction
Exosomes in Urine: Differences in Gene Expression | just before end of surgery
  - Gene expression and expression comparison in exosomes The gene expression difference is determined using the SAM tool and DEseq2, and the Gene Ontology (GO) Database (www.geneontology.org) and the KEGG database (www.genome.jp/kegg) are used to find the correlation between gene functions.
  In the case of miRNA, there will be a regulatory function of the coding gene, so for this purpose, an integrative analysis is performed to identify the mRNA-miRNA interaction
Exosomes in Urine: Differences in Gene Expression | Post operative day 1 (6 AM)
  - Gene expression and expression comparison in exosomes The gene expression difference is determined using the SAM tool and DEseq2, and the Gene Ontology (GO) Database (www.geneontology.org) and the KEGG database (www.genome.jp/kegg) are used to find the correlation between gene functions.
  In the case of miRNA, there will be a regulatory function of the coding gene, so for this purpose, an integrative analysis is performed to identify the mRNA-miRNA interaction
Exosomes in Urine: Differences in Gene Expression | Post operative day 1 (6 PM)
  - Gene expression and expression comparison in exosomes The gene expression difference is determined using the SAM tool and DEseq2, and the Gene Ontology (GO) Database (www.geneontology.org) and the KEGG database (www.genome.jp/kegg) are used to find the correlation between gene functions.
  In the case of miRNA, there will be a regulatory function of the coding gene, so for this purpose, an integrative analysis is performed to identify the mRNA-miRNA interaction
Exosomes in Urine: Differences in Gene Expression | immediately after onset of delirium
  - Gene expression and expression comparison in exosomes The gene expression difference is determined using the SAM tool and DEseq2, and the Gene Ontology (GO) Database (www.geneontology.org) and the KEGG database (www.genome.jp/kegg) are used to find the correlation between gene functions.
  In the case of miRNA, there will be a regulatory function of the coding gene, so for this purpose, an integrative analysis is performed to identify the mRNA-miRNA interaction
Exosomes in Urine: Differences in Gene Expression | 7 days after surgery, within hospitalization period
  - Gene expression and expression comparison in exosomes The gene expression difference is determined using the SAM tool and DEseq2, and the Gene Ontology (GO) Database (www.geneontology.org) and the KEGG database (www.genome.jp/kegg) are used to find the correlation between gene functions.
  In the case of miRNA, there will be a regulatory function of the coding gene, so for this purpose, an integrative analysis is performed to identify the mRNA-miRNA interaction
Exosomes in Blood: Differences in Gene Expression | Just before surgery
  - Gene expression and expression comparison in exosomes The gene expression difference is determined using the SAM tool and DEseq2, and the Gene Ontology (GO) Database (www.geneontology.org) and the KEGG database (www.genome.jp/kegg) are used to find the correlation between gene functions.
  In the case of miRNA, there will be a regulatory function of the coding gene, so for this purpose, an integrative analysis is performed to identify the mRNA-miRNA interaction
Exosomes in Blood: Differences in Gene Expression | just before end of surgery
  - Gene expression and expression comparison in exosomes The gene expression difference is determined using the SAM tool and DEseq2, and the Gene Ontology (GO) Database (www.geneontology.org) and the KEGG database (www.genome.jp/kegg) are used to find the correlation between gene functions.
  In the case of miRNA, there will be a regulatory function of the coding gene, so for this purpose, an integrative analysis is performed to identify the mRNA-miRNA interaction
Fecal microbiota | just before surgery, on the day of discharge

SECONDARY OUTCOMES:
Brain efficiency test(EEG) | Before surgery (from 2 weeks before to the day before)
  - EEG test for brain efficiency Peak-MEF(intermediate rhythm of background EEG spectrum), Peak-Freq, Peak_power, Theta frequency band (4 or more and less than 8) of the left (Fp1) EEG power value (log scale), Left (Fp1) EEG alpha frequency band (8 or more and less than 12) Power value (log scale), Left (Fp1) EEG slow beta band (more than 12 and less than 15) power value (log scale), Left (Fp1) EEG mid-beta frequency band (more than 15 and less than 20) power value (log scale), Fast beta frequency band of the left (Fp1) brain waves (more than 20 and less than 30) power value (log scale), Gamma frequency band (30 or more and 50 or less) power value (log scale) of left (Fp1) brain waves, Peak amplitude of 125 Hz auditory stimulated brain potential (ERP); Left and right average of P2 (maximum) peak value difference based on N1 (minimum) peak. Peak amplitude mean of left (Fp1) auditory induced brain potentials (ERPs), Left and right EEG cross-correlation coefficient.
Brain efficiency test(pulse wave test) | Before surgery (from 2 weeks before to the day before)
  - pulse wave test for brain efficiency HF (High Frequency) frequency band of heart rate variability (RRV) (0.15 or more and 0.4Hz or less), LF (Low Frequency) frequency band of heart rate variability (RRV) (0.04 or more and less than 0.15 Hz) absolute power, Relative percentage of LF to (LF + HF), Total power of heart rate variability (RRV), Heart rate variability (RRV) histogram; the histogram distribution area divided by the maximum value
Cognitive test -MMSE | Before surgery (from 2 weeks before to the day before)
Cognitive test -MOCA | Before surgery (from 2 weeks before to the day before)
Cognitive test -TICS | Before surgery (from 2 weeks before to the day before)
Brain efficiency test(EEG) | 7 days after surgery, within hospitalization period
  - EEG test for brain efficiency Peak-MEF(intermediate rhythm of background EEG spectrum), Peak-Freq, Peak_power, Theta frequency band (4 or more and less than 8) of the left (Fp1) EEG power value (log scale), Left (Fp1) EEG alpha frequency band (8 or more and less than 12) Power value (log scale), Left (Fp1) EEG slow beta band (more than 12 and less than 15) power value (log scale), Left (Fp1) EEG mid-beta frequency band (more than 15 and less than 20) power value (log scale), Fast beta frequency band of the left (Fp1) brain waves (more than 20 and less than 30) power value (log scale), Gamma frequency band (30 or more and 50 or less) power value (log scale) of left (Fp1) brain waves, Peak amplitude of 125 Hz auditory stimulated brain potential (ERP); Left and right average of P2 (maximum) peak value difference based on N1 (minimum) peak. Peak amplitude mean of left (Fp1) auditory induced brain potentials (ERPs), Left and right EEG cross-correlation coefficient.
Brain efficiency test(pulse wave test) | 7 days after surgery, within hospitalization period
  - pulse wave test for brain efficiency HF (High Frequency) frequency band of heart rate variability (RRV) (0.15 or more and 0.4Hz or less), LF (Low Frequency) frequency band of heart rate variability (RRV) (0.04 or more and less than 0.15 Hz) absolute power, Relative percentage of LF to (LF + HF), Total power of heart rate variability (RRV), Heart rate variability (RRV) histogram; the histogram distribution area divided by the maximum value
Cognitive test -MMSE | 7 days after surgery, within hospitalization period
Cognitive test -MOCA | 7 days after surgery, within hospitalization period
Cognitive test -TICS | 7 days after surgery, within hospitalization period
Brain efficiency test(EEG) | 1 month after surgery
  - EEG test for brain efficiency Peak-MEF(intermediate rhythm of background EEG spectrum), Peak-Freq, Peak_power, Theta frequency band (4 or more and less than 8) of the left (Fp1) EEG power value (log scale), Left (Fp1) EEG alpha frequency band (8 or more and less than 12) Power value (log scale), Left (Fp1) EEG slow beta band (more than 12 and less than 15) power value (log scale), Left (Fp1) EEG mid-beta frequency band (more than 15 and less than 20) power value (log scale), Fast beta frequency band of the left (Fp1) brain waves (more than 20 and less than 30) power value (log scale), Gamma frequency band (30 or more and 50 or less) power value (log scale) of left (Fp1) brain waves, Peak amplitude of 125 Hz auditory stimulated brain potential (ERP); Left and right average of P2 (maximum) peak value difference based on N1 (minimum) peak. Peak amplitude mean of left (Fp1) auditory induced brain potentials (ERPs), Left and right EEG cross-correlation coefficient.
Brain efficiency test(pulse wave test) | 1 month after surgery
  - pulse wave test for brain efficiency HF (High Frequency) frequency band of heart rate variability (RRV) (0.15 or more and 0.4Hz or less), LF (Low Frequency) frequency band of heart rate variability (RRV) (0.04 or more and less than 0.15 Hz) absolute power, Relative percentage of LF to (LF + HF), Total power of heart rate variability (RRV), Heart rate variability (RRV) histogram; the histogram distribution area divided by the maximum value
Cognitive test -MMSE | 1 month after surgery
Cognitive test -MOCA | 1 month after surgery
Cognitive test -TICS | 1 month after surgery
Brain efficiency test(EEG) | 1 year after surgery
  - EEG test for brain efficiency Peak-MEF(intermediate rhythm of background EEG spectrum), Peak-Freq, Peak_power, Theta frequency band (4 or more and less than 8) of the left (Fp1) EEG power value (log scale), Left (Fp1) EEG alpha frequency band (8 or more and less than 12) Power value (log scale), Left (Fp1) EEG slow beta band (more than 12 and less than 15) power value (log scale), Left (Fp1) EEG mid-beta frequency band (more than 15 and less than 20) power value (log scale), Fast beta frequency band of the left (Fp1) brain waves (more than 20 and less than 30) power value (log scale), Gamma frequency band (30 or more and 50 or less) power value (log scale) of left (Fp1) brain waves, Peak amplitude of 125 Hz auditory stimulated brain potential (ERP); Left and right average of P2 (maximum) peak value difference based on N1 (minimum) peak. Peak amplitude mean of left (Fp1) auditory induced brain potentials (ERPs), Left and right EEG cross-correlation coefficient.
Brain efficiency test(pulse wave test) | 1 year after surgery
  - pulse wave test for brain efficiency HF (High Frequency) frequency band of heart rate variability (RRV) (0.15 or more and 0.4Hz or less), LF (Low Frequency) frequency band of heart rate variability (RRV) (0.04 or more and less than 0.15 Hz) absolute power, Relative percentage of LF to (LF + HF), Total power of heart rate variability (RRV), Heart rate variability (RRV) histogram; the histogram distribution area divided by the maximum value
Cognitive test -MMSE | 1 year after surgery
Cognitive test -MOCA | 1 year after surgery
Cognitive test -TICS | 1 year after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No